CLINICAL TRIAL: NCT02545985
Title: Novel Sirolimus-eluting Stent Prolim® With a Biodegradable Polymer in the All-comers Population
Brief Title: First-in-man Sirolimus-eluting Prolim® Stent Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Jacek Bil, MD, PhD, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2015-08-30; First posted 2015-09-10 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Sirolimus-eluting Stainless Steel Coronary Stent Prolim®
Keywords: sirolimus; coronary stent; Prolim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prolim stent implantation (Experimental): In patients with symptomatic coronary artery disease Prolim stent was implanted in coronary arteries
  Interventions: Device: Prolim stent deployment

INTERVENTIONS:
Device: Prolim stent deployment — Prolim stent was implanted in patients who signed the informed consent and met the exclusion and inclusion criteria.

SUMMARY:
The aim of this study was to assess the safety and the efficacy of the novel sirolimus-eluting Prolim® stent with a biodegradable polymer in the all-comers population.

DETAILED DESCRIPTION:
Investigators prospectively enrolled all patients with stable coronary artery disease or acute coronary syndrome, treated with Prolim® stent between January and December 2013 in two interventional cardiology centers in Poland. Angiographic control was planned at 12 months, in which 15% of patients (randomly chosen) underwent optical coherence tomography analysis. The primary end-point was the cumulative rate of cardiac death, myocardial infarction, and target lesion revascularization after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old,
* stable coronary artery disease (SCAD) or acute coronary syndrome (unstable angina - UA, non-ST elevation myocardial infarction - NSTEMI or ST-elevation myocardial infarction - STEMI) and
* signed informed consent

Exclusion Criteria:

* inability to take dual antiplatelet therapy for 12 months,
* left ventricular ejection fraction ≤ 30%,
* chronic total occlusions, and
* in-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the cumulative rate of major adverse cardiovascular events (MACE). | 12 months
  consisting of cardiac death, myocardial infarction (MI) and clinically-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Secondary endpoints included the rates of cardiac death, all-cause death, MI, TLR, TVR and stent thrombosis. | 12 moths
  Secondary endpoints included the rates of cardiac death, all-cause death, MI, TLR, TVR and stent thrombosis.
Late lumen loss (LLL) | 12 moths
  The value (in mm) of LLL assessed in qualitative coronary angiography (QCA)
The percentage of covered struts assessed in optical coherence tomography (OCT) | 12 months
  The percentage of covered struts assessed in OCT
The neointima volume assessed in OCT | 12 months
  The neointima volume (in mm3) assessed in OCT
The device success rate | intraoperative
  The percentage of Prolim stents successfully implanted.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Bil, MD, PhD, Principal Investigator — Central Clinical Hospital of the Ministry of Internal Affairs

REFERENCES:
- [Result] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Result] Lavi S, Dzavik V. Biodegradable Stent Platforms: Are We Heading in the Right Direction? Can J Cardiol. 2015 Aug;31(8):957-9. doi: 10.1016/j.cjca.2015.04.005. Epub 2015 Apr 14. No abstract available. PMID 26095938
- [Result] Nagoshi R, Shinke T, Otake H, Shite J, Matsumoto D, Kawamori H, Nakagawa M, Kozuki A, Hariki H, Inoue T, Ohsue T, Taniguchi Y, Iwasaki M, Nishio R, Hiranuma N, Konishi A, Kinutani H, Miyoshi N, Takaya T, Yamada S, Yasaka Y, Hayashi T, Yokoyama M, Kato H, Kadotani M, Ohnishi Y, Hirata K. Qualitative and quantitative assessment of stent restenosis by optical coherence tomography: comparison between drug-eluting and bare-metal stents. Circ J. 2013;77(3):652-60. doi: 10.1253/circj.cj-12-0610. Epub 2012 Dec 21. PMID 23257388
- [Result] Zhang Q, Qiu JP, Kirtane AJ, Zhu TQ, Zhang RY, Yang ZK, Hu J, Ding FH, DU R, Shen WF. Comparison of biodegradable polymer versus durable polymer sirolimus-eluting stenting in patients with acute st-elevation myocardial infarction undergoing primary percutaneous coronary intervention: results of the RESOLVE study. J Interv Cardiol. 2014 Apr;27(2):131-41. doi: 10.1111/joic.12102. PMID 24697948
- [Derived] Bil J, Gil RJ, Kern A, Pawlowski T, Seweryniak P, Sliwinski Z. Novel sirolimus-eluting stent Prolim(R) with a biodegradable polymer in the all-comers population: one year clinical results with quantitative coronary angiography and optical coherence tomography analysis. BMC Cardiovasc Disord. 2015 Nov 14;15:150. doi: 10.1186/s12872-015-0139-5. PMID 26573577